CLINICAL TRIAL: NCT01859559
Title: A Randomized Controlled Trial To Compare The Initial Success Rate of Ultrasound Guided Versus Landmark Approach For Placement of Peripheral Intravenous Access Lines in Emergency Department Patients
Brief Title: Evaluate Initial Success Rate of Ultrasound Guided Versus Landmark Approach For Peripheral Intravenous Access
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Melissa McCarthy, Associate Professor, George Washington University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIV-RCT-ED
Record Dates: First submitted 2013-05-16; First posted 2013-05-22 (Estimated); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Patients With Peripheral Intravenous Access Lines
Keywords: ultrasound; peripheral intravenous access; operator experience

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Easy Access (Experimental): This arm will included emergency department patients that are judged to have easy intravenous access in at least one of the upper extremities by the ED technician.
  Interventions: Procedure: Ultrasound-guided peripheral intravenous access line placement; Procedure: Landmark Approach to peripheral intravenous access line placement
- Difficult Access By Clinician Judgment (Experimental): This arm will include patients that at least one vein is visible or palpable in one of the upper extremities but either the ED technician and/or ED nurse judges the patient to have difficult intravenous access.
  Interventions: Procedure: Ultrasound-guided peripheral intravenous access line placement; Procedure: Landmark Approach to peripheral intravenous access line placement
- Non visible and Non palpable (Experimental): This arm will include patients for whom neither the ED technician nor an ED nurse can identify a visible or palpable vein that is suitable for an intravenous access line in either upper extremity.
  Interventions: Procedure: Ultrasound-guided peripheral intravenous access line placement; Procedure: Landmark Approach to peripheral intravenous access line placement

INTERVENTIONS:
Procedure: Ultrasound-guided peripheral intravenous access line placement — The ED technician will use an ultrasound machine with a vascular probe to visualize the vein and guide the PIV line using a one-operator dynamic technique.
Procedure: Landmark Approach to peripheral intravenous access line placement — ED technician will use standard anatomical landmarks and palpation to puncture the skin and insert the peripheral intravenous access line in the upper extremity.

SUMMARY:
The primary objective of this randomized controlled trial (RCT) is to compare the success rate of obtaining peripheral vascular access with ultrasound guidance versus the traditional, landmark approach among patients with varying degrees of intravenous access difficulty. In addition to comparing overall initial success rates of the two methods, we will also compare the success rates by degree of intravenous access difficulty (3 main subject subgroups) and by operator experience (approximately 20 emergency department technicians).

The main hypothesis is that the initial success rate will be significantly higher (5% or greater) for ultrasound guided peripheral intravenous access compared to landmark approach among patients who are judged to have difficult intravenous access but no significant difference (i.e. < 5%) among patients judged to have easy intravenous access.

DETAILED DESCRIPTION:
This is a randomized controlled trial with a two group parallel design that will compare the initial success rate of peripheral intravenous line (PIV) placement between the traditional, landmark approach versus ultrasound guided. Emergency department (ED) patients who are in a treatment room and require a PIV line are eligible for the study. For those who are eligible, the ED technician and an ED nurse will each complete a clinical data sheet that documents the degree of IV access difficulty.

For those who enroll, the research assistant (RA) will randomize the subject to one of two treatment groups: (1) ultrasound guided or; (2) landmark approach. The ED technician will perform the PIV placement based on the treatment group assigned through the randomization process. The RA will be present during the PIV placement and will ask the patient prior to the procedure about factors that may influence IV access (i.e. self-reported weight and height, presence of chronic conditions). The RA will also document the ED outcomes of the procedure (i.e. duration of procedure, success or failure, complications of procedure) and query the patient on the extent of discomfort associated with the procedure. Finally, for those subjects who are admitted to the hospital, a RA will conduct follow-up on the PIV line to determine how long it is used on the ward and the reason for taking it out (i.e. no longer needed, infection, infiltration, fell out, etc). It is hospital policy that PIV lines be changed every 72 hours to prevent infection so we anticipate that the maximum follow-up of each ED PIV line placed will be 72 hours.

There are two treatment groups, the ultrasound guided treatment group and the traditional, landmark group. For both treatment groups, a tourniquet will be placed above the upper extremity vein chosen for cannulation. For the landmark approach, the ED technician will use standard anatomical landmarks and palpation to puncture the skin and insert the IV line. If the patient is randomized to the ultrasound group, the operator will use ultrasound to help visualize the vein and direct line placement. When using ultrasound, the ED technicians will employ a one-person technique. For both treatment groups, if the first attempt fails, we will randomize the subject again to one of the two treatment arms. We are randomizing a second time because failure at first attempt is a good marker of the difficulty of the procedure. By randomizing a second time, we will be able to determine whether either method is superior after one failed attempt. After the second failed attempt, the ED technician can use whatever method he/she chooses to place the line.

Because of the nature of the intervention, this RCT is unblinded.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* peripheral venous (PIV) access line ordered by a physician during their emergency department visit.

Exclusion Criteria:

* Non-English or non-spanish speaking
* already enrolled in a different study during the ED visit
* too sick, patient requires intravenous access quickly and can not take the time to enroll in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1189 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Initial success rate | immediatetely after first attempt, average attempt takes 15 minutes
  A successful cannulation (blood return or ability to infuse intravenous fluid without infiltration) on initial percutaneous needle puncture.

SECONDARY OUTCOMES:
Any complications associated with the PIV line | within ED visit, average ED length of stay is 6 hours
  Incidence of infiltration, arterial puncture, or nerve puncture

OTHER OUTCOMES:
Numeric Rating of Pain Associated with insertion of PIV line | within 5 minutes of final PIV placement, average placement take < 30 minutes
  Patient-reported measure of pain associated with the insertion of the PIV line using the Numeric Rating Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa L McCarthy, ScD, Principal Investigator — George Washington University; Hamid Shokoohi, MD, Principal Investigator — George Washington University
Locations (1):
- George Washington University Hospital, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Heinrichs J, Fritze Z, Vandermeer B, Klassen T, Curtis S. Ultrasonographically guided peripheral intravenous cannulation of children and adults: a systematic review and meta-analysis. Ann Emerg Med. 2013 Apr;61(4):444-454.e1. doi: 10.1016/j.annemergmed.2012.11.014. Epub 2013 Feb 15. PMID 23415740
- [Background] McCarthy ML, Shokoohi H, Boniface KS, Eggelton R, Lowey A, Lim K, Shesser R, Li X, Zeger SL. Ultrasonography Versus Landmark for Peripheral Intravenous Cannulation: A Randomized Controlled Trial. Ann Emerg Med. 2016 Jul;68(1):10-8. doi: 10.1016/j.annemergmed.2015.09.009. Epub 2015 Oct 23. PMID 26475248
- [Derived] Shokoohi H, Boniface KS, Kulie P, Long A, McCarthy M. The Utility and Survivorship of Peripheral Intravenous Catheters Inserted in the Emergency Department. Ann Emerg Med. 2019 Sep;74(3):381-390. doi: 10.1016/j.annemergmed.2019.02.003. Epub 2019 Mar 27. PMID 30926188